CLINICAL TRIAL: NCT00656825
Title: Multicentre, Placebo-Controlled, Multi-Dosis, Phase I Clinical Trial to Evaluate the Tolerability and Bioavailability of TGF β1 Inhibitor Peptide 144 After Topical Administration in Healthy Volunteers.
Brief Title: Tolerability and Bioavailability of the P144 Peptide Inhibitor of TGF-β1 After Topical Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ISDIN (Industry)
Collaborators: Digna Biotech S.L. (Industry)
Responsible Party: ISDIN, ISDIN
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NAFB001-SS-01; 2006-002755-33
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Healthy
Keywords: P144; TGF-β1; Healthy volunteers; Cutaneous tolerability; Skin fibrosis; systemic scleroderma; systemic sclerosis; Safety
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Panel I (Active Comparator): The first 12 subjects will be selected and ranodmized in order to receive the first treatment dose of 100 μg/mL or placebo in a 8:4 ratio
  Interventions: Drug: P144 cream
- Panel II (Active Comparator): The second 12 subjects will be selected and randomized in order to receive the second treatment dose of 200 μg/mL or placebo in a 8:4 ratio
  Interventions: Drug: P144 cream
- Panel III (Active Comparator): The third 12 subjects will be selected and randomized in order to receive the third treatment dose of 300 μg/mL or placebo in a 8:4 ratio
  Interventions: Drug: P144 cream
- Placebo (Placebo Comparator): Patients from each panel will be given placebo in a 4:8 ratio.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: P144 cream — P144 cream will be given at a dose of 100 μg/mL
  Arms: Panel I
Drug: P144 cream — P144 cream will be given at a dose of 200 μg/mL
  Arms: Panel II
Drug: P144 cream — P144 cream will be given at a dose of 300 μg/mL
  Arms: Panel III
Drug: Placebo — Placebo will be randomly given to 4 subjects in each panel
  Arms: Placebo

SUMMARY:
Transforming growth factor-beta 1 (TGF-β1) is consistently over expressed in most fibrotic diseases and displays a variety of profibrotic effects in fibroblasts. Activation of TGF-β receptors induces the activation of several kinase signalling cascades leading to the phosphorylation of SMAD proteins as well as to the activation of SMAD-independent kinases that collectively activate ECM synthesis and fibroblast growth and differentiation into myofibroblasts. TGF-β1 is one of the main mediators in the fibrotic process, associated to both scarring and a long list of pathologies related to chronic inflammation and which affect all type of organs and tissues. An increase in TGF-β1 mRNA and protein levels has been described in these processes. Peptide 144 (P144) is the acetic salt of a 14mer peptide from human TGF-β1 type III receptor (betaglycan). P144 TGF-β1-inhibitor has been specifically designed to block the interaction between TGF-β1 and TGF-β1 type III receptor, thus blocking its biological effects. P144 has shown significant antifibrotic activity in mice receiving repeated subcutaneous injections of bleomycin, a widely accepted animal model of human scleroderma, and could contribute to the development. The purpose of this study is to assess the tolerability and safety of topical application of P144 in healthy volunteers.

DETAILED DESCRIPTION:
Three different formulations of DIGNA P144 cream (containing 100 μg/mL, 200 μg/mL and 300 μg/mL) will be tested in healthy volunteers. Tolerability evaluation is performed through the specific cutaneous tolerability visual scale of Frosch and Kligman. Safety assessment is carried out by studying vital signs, physical examination, by performing laboratory tests, electrocardiogram and reporting any adverse events experienced. This is the first time that P144 will be administered in humans. The topical route has been chosen since the indication for which P144 is going to be clinically developed will be cutaneous sclerosis associated to scleroderma.

Systemic sclerosis or scleroderma is a multisystemic disorder characterized by the excessive synthesis and deposition of extracellular matrix proteins that result in the fibrosis of skin and visceral organs (including gastrointestinal tract, lungs, heart and kidneys).

The pathogenesis of scleroderma is complex and still poorly understood, but major pathways involved in the development of the condition are microvascular and immunological abnormalities, as well as dysregulation of fibroblast activity. One of the key molecules involved in the pathogenesis of skin fibrosis is the TGF-β1; TGF-β1 is a cytokine directly responsible for fibroblasts proliferation and collagen and extracellular matrix overproduction.

The affected skin of patients with systemic sclerosis gradually becomes firm, thickened and eventually tightly bound to underlying subcutaneous tissue (indurative phase). It loses hair, oil, and sweat glands becoming dry and coarse. Changes begin distally in the extremities and advance proximally. Lesions develop over a period of time varying from months to a few years. In patients with limited scleroderma, only the skin of fingers, hands, face and lower arms and legs is affected. On the contrary, patients with the diffuse cutaneous disease, skin changes will become generalized, involving initially the extremities and followed by the face and trunk. Rapid progression of these changes over a 2 to 3 year period is usually associated with a greater risk of visceral disease. After several years of disease, the skin may soften and return to normal thickness or become thin and atrophic.

There is currently no approved specific treatment for skin fibrosis in systemic sclerosis neither in the European Union nor the United States of America. P144 belongs to a peptide family that is able to inhibit TGF-β1 in both in vitro and in vivo models characterized by excessive TGF-β1 function. Topical application of P144 exerts a preventive effect precluding the induction of skin fibrosis and the accumulation of collagen in these animals and also has shown its therapeutic properties reducing the skin fibrosis and soluble collagen content in mice with established fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol specific procedures are performed.
* Age between 18 and 45 years old
* Skin phenotype I to IV following Fitzpatrick's classification scale
* BMI between 20-29 kg/sqm
* Not clinically relevant alterations in: arterial pressure, cardiac frequency, analytical values (Hematology, Biochemistry, Urianalysis, Coagulation, Serology, Toxics)

Exclusion Criteria:

* Pregnany or lactancy
* Allergy to any medication
* Subjects with skin illnesses or systemic illnesses with skin afectation
* History of drug abuse or regular consumption of alcohol
* Participation in other clinical trials 3 months before the signature of the informed consent
* UV exposure or sun exposure on the zone to be treated
* History of skin hypersensitivity
* Chronic treatment with anti-inflammatories or anti-histaminics
* Treatment with corticoids on the previous month
* Hyperpigmentation on the zone to be treated

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Tolerability evaluation was performed through the specific cutaneous tolerability visual scale of Frosch and Kligman. | Twenty-one days

SECONDARY OUTCOMES:
Safety assessment was carried out by studying vital signs, physical examination, by performing laboratory tests, electrocardiogram and reporting any adverse events experienced. Bioavailability of P 144 in serum. | Twenty-one days

CONTACTS AND LOCATIONS:
Overall Officials: Belén Ruiz, MD, Principal Investigator — Hospital Universitario Puerta de Hierro; Belén Sádaba, MD, Principal Investigator — Clínica Universitaria de Navarra
Locations (2):
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Madrid, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Pamplona